CLINICAL TRIAL: NCT00252564
Title: Randomized PhIII Trial of Cetuximab, Bevacizumab & Biweekly Infusional 5FU/Leucovorin (FOLF-CB) vs. Oxaliplatin, Bevacizumab, & Biweekly Infusional 5FU/Leucovorin (Bev-FOLFOX) in First Line Treatment of Metastatic Colorectal Cancer
Brief Title: Cetuximab, Bevacizumab & 5FU/Leucovorin vs. Oxaliplatin, Bevacizumab & 5FU/Leucovorin in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Memorial Sloan Kettering Cancer Center (Other); Prologue Research International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-041
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bev-FOLFOX (Experimental): (Bev-FOLFOX): Bevacizumab, followed by oxaliplatin and LV given simultaneously via "T" connector over 2 hours, followed by bolus 5-FU followed by infusional 5-FU.
  Bevacizumab --> oxaliplatin and LV --> bolus 5-FU --> infusional 5-FU
  Dosing on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- FOLF-CB (Experimental): (FOLF-CB): Cetuximab administered over 2 hours (first dose only; administer all other doses over 1 hour) followed by bevacizumab over 30 minutes, followed by LV over 30 minutes, followed by bolus 5-FU followed by infusional 5-FU.
  Cetuximab --> bevacizumab --> LV --> bolus 5-FU --> infusional 5-FU
  Interventions: Drug: Bevacizumab; Drug: Leucovorin; Drug: Fluorouracil; Drug: Cetuximab

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg over 30 minutes on Days 1 and 15
  Other Names: Avastin
Drug: Oxaliplatin — 85 mg/m2 on Days 1 and 15
  Other Names: Eloxatin
  Arms: Bev-FOLFOX
Drug: Leucovorin — 400 mg/m2 on Days 1 and 15
Drug: Fluorouracil — 400 mg/m2, IV bolus followed by: 1200 mg/m2/day via 24-hour continuous infusion, for 2 consecutive days (total 5-FU infusion dose = 2400 mg/m2 over the 48 hour period)
  Other Names: 5FU
Drug: Cetuximab — 400 mg/m2 over 2 hours (Cycle 1 Day 1 only) All subsequent doses (Day 8, 15, 22 of Cycle 1 and Days 1, 8, 15, 22 other cycles)250 mg/m2 over 1 hour
  Other Names: Erbitux
  Arms: FOLF-CB

SUMMARY:
The purpose of this study is to compare the rates of Progression-Free Survival (PFS) at 12 months for patients treated with Bev-FOLFOX versus patients treated with FOLF-CB for first line treatment of metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a Phase III, open label, nonblinded study. A total of 240 eligible patients will be randomized on a 1:1 basis to either treatment Arm.

In this trial, we will compare the efficacy, safety, and tolerability of this novel combination of biweekly infusional 5-FU/leucovorin plus cetuximab and bevacizumab (FOLF-CB) to the current standard of care, biweekly infusional 5-FU/leucovorin plus oxaliplatin and bevacizumab (Bev-FOLFOX). For practical purposes, this study will be a head to head comparison of oxaliplatin versus cetuximab, since the other components of both regimens will be the same.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically or cytologically confirmed colorectal cancer with metastatic disease
* Measurable disease
* Previously irradiated lesions will be considered evaluable, if they progressed since radiation
* Has disease other than limited to surgically resectable liver-only or lung-only metastatic disease
* Not received prior chemo and/or biotherapy for metastatic disease
* Not received oxaliplatin, bevacizumab, or cetuximab in the adjuvant setting
* May have received 5-FU, leucovorin, and/or irinotecan in the adjuvant setting, however must have remained free of disease recurrence (including free of abnormal CEA level) for 1- year or more
* Is >18 years of age
* ECOG performance status 0 or 1
* Normal organ & marrow function
* Use of an acceptable method of birth control
* Not pregnant or breast feeding
* Paraffin tissue block(s) or 12 (minimum) unstained slides available, for assessment of potential predictive markers related to the EGFR, VEGF, DNA repair, and fluoropyrimidine catabolism pathways. If no block is available, slides (typically 7 to 10 um sections, air dried on uncharged slides) may be sent
* Signed a Patient Informed Consent Form
* Signed a Patient Authorization Form (HIPAA) Form

EXCLUSION CRITERIA:

* Had prior chemotherapy for metastatic colorectal cancer
* Received any prior treatment with oxaliplatin, bevacizumab, or cetuximab in the adjuvant treatment of their colorectal cancer
* Currently receiving any other investigational anticancer agents or has participated in an experimental drug study within the past 4 weeks
* History of primary CNS tumors, seizures not well-controlled with standard medical therapy, or stroke
* Sustained hypertension, as characterized by persistent blood pressures greater than 150/100 despite medical management
* New York Heart Association (NYHA) Grade II or greater congestive heart failure or has had angioplasty or placement of coronary stents within the past 6 months
* Clinically significant peripheral vascular disease
* History of serious allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, cetuximab, oxaliplatin, fluorouracil, leucovorin, or other agents used in the study
* Received prior cetuximab or other EGFR-directed therapy, or history of prior anti-cancer murine or chimeric monoclonal antibody therapy; prior humanized and human monoclonal antibody therapy is also excluded.
* Received prior treatment with bevacizumab or other agents specifically targeting VEGF or VEGF receptors
* Uncontrolled intercurrent illness including, not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the Investigator/Treating Physician
* Serious or non-healing active wound ulcer, or active bone fracture
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of protocol treatment
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 1
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Current or recent use of a thrombolytic agent within last 30 days. Use for clearance of central line catheter is permitted.
* Evidence of bleeding diathesis (disorder) or clinically significant coagulopathy (Note that deep venous thrombosis is not regarded as a reason for exclusion from this trial)
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of arterial thromboembolic events within 6 months
* Urine protein:creatinine ratio greater than 1.0 at screening
* Pregnant or lactating woman
* Known to be HIV positive or receiving combination anti-retroviral therapy
* Unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Cohn, MD, Principal Investigator — US Oncology Research; Leonard Saltz, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (81):
- United States (81):
  - Brimingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Assoc, Sedona, Arizona
  - Business Office - ACRC, Tucson, Arizona
  - Cancer Care Associates of Fresno Medical Group, Inc (aka California Cancer Care), Fresno, California
  - Monterey Bay Oncology, Monterey, California
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Greeley Medical Clinic Oncology Hematology, PC, Greeley, Colorado
  - Connecticut Oncology & Hematology, LLP, Torrington, Connecticut
  - Integrated Community Oncology Network (ICON) / fka:Florida Oncology Associates, Jacksonville, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Medical Oncology Associates of Augusta PC, Augusta, Georgia
  - Spalding Oncology Services, Griffin, Georgia
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Fort Wayne Medical Oncology Hematology, Inc, Fort Wayne, Indiana
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Auerbach Hematology Oncology Associated, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Osteopathic Medical Oncology and Hematology, Clinton Township, Michigan
  - Kalamazoo Hematology & Oncology, Kalamazoo, Michigan
  - Hematology Oncology Associates of Ohio & Michigan, Lambertville, Michigan
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Centers, Las Vegas, Nevada
  - Hematology-Oncology Associates of NNJ, PA, Morristown, New Jersey
  - New York Oncology Hematology, PC, Albany, New York
  - North Shore Hematology, East Setauket, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Northwestern Carolina Ocology Hemato, Hickory, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Cancer Center Associates of Carolina, PA / fka Carolina Cancer Center, Aiken, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - C. Michael Jones, MD, Germantown, Tennessee
  - Texas Cancer Center-Abilene (Shouth), Abilene, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, PA - Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - Texas Cancer Center-Denton, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - San Antonio Tumor & Blood Clinic, Fredericksburg, Texas
  - Texas Oncology, PA, Garland, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - HOAST - Medical Dr., San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care and Research Center, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Texas Oncology, PA, Webster, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Puget Sound Cancer Center Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley mem Hosp/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 247 patients were recruited from multiple research sites and were randomly assigned to either Arm A or Arm B between December 2005 to June 2007.
Pre-assignment Details: The patients were required to be in screening for up to 3 weeks prior to registering the patient for randomization
Groups:
- Arm A: (Bev-FOLFOX): Bevacizumab, followed by oxaliplatin and LV given simultaneously via "T" connector over 2 hours, followed by bolus 5-FU followed by infusional 5-FU.
  Bevacizumab --> oxaliplatin and LV --> bolus 5-FU --> infusional 5-FU
  Dosing on Days 1 and 15 of each 28-day cycle
- Arm B: (FOLF-CB): Cetuximab administered over 2 hours (first dose only; administer all other doses over 1 hour) followed by bevacizumab over 30 minutes, followed by LV over 30 minutes, followed by bolus 5-FU followed by infusional 5-FU.
  Cetuximab --> bevacizumab --> LV --> bolus 5-FU --> infusional 5-FU
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 124 (From randomization) | 123 (From randomization)
Completed | 85 (Received 6+ cycles OR had response (RECIST criteria, CR or PR)) | 79 (Received 6+ cycles OR had response (RECIST criteria, CR or PR))
Not Completed | 39 | 44
Not completed — Adverse Event | 17 | 13
Not completed — Unrelated Complication | 2 | 1
Not completed — Disease Progression | 14 | 20
Not completed — Death | 0 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Patient Request | 4 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 67 | 140
  >=65 years | 51 | 56 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 63 (11) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 104
  Male | 70 | 73 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 100 | 99 | 199
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 124 | 123 | 247

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: From randomization to first progression or death, whichever comes first (event); or first new anti-cancer treatment if before or without progression / death (censoring); or last follow-up date otherwise (censoring).
  Kaplan-Meier median PFS time and PFS rate (at 12 months)
Time Frame: 12 months
Population: This analysis included all registered (or randomized) patients, i.e. intent-to-treat (ITT) population, regardless of patient's treatment status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 124 | 123
months | 11.0 [9.2 to 13.6] | 8.3 [6.7 to 9.7]

2. Primary Outcome: Progression-free Survival (PFS) Rate at 1 Year.
Description: From randomization to first progression or death, whichever comes first (event); or first new anti-cancer treatment if before or without progression / death (censoring); or last follow-up date otherwise (censoring).
Time Frame: 12 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: proportion of participants w/ PFS at 1yr
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 124 | 123
proportion of participants w/ PFS at 1yr | 0.45 [0.34 to 0.55] | 0.32 [0.23 to 0.42]

3. Secondary Outcome: Overall Survival (OS)
Description: From randomization to death (event); or last follow-up date if alive (censoring).
  Kaplan-Meier OS median time.
Time Frame: up to 4 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 124 | 123
Months | 21.3 [18.2 to 25.2] | 19.5 [16.5 to 21.6]

4. Secondary Outcome: Objective Response Rate
Description: Percentage of patients with tumor response (by RECIST criteria, including complete response, or CR, i.e. disappearance of all target lesions; and partial response, or PR, i.e. at least a 30% decrease in the sum of the longest diameters of target lesions taking as reference the baseline sum of the longest diameters) among all "per-protocol population" patients.
Time Frame: 12 months
Population: This analysis included all eligible and treated patients, i.e. per-protocol population. A patient will be considered in the arm he/she is actually treated, not randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 117 | 119
percentage of participants | 52.1 [42.7 to 61.5] | 41.2 [32.2 to 50.6]

ADVERSE EVENTS:
Time Frame: during the whole treatment period, up to 30 days following last dose
Description: for treated patients only, assessed at each treatment visit
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 40/118 | 49/121
Other Adverse Events (participants affected / at risk) | 117/118 | 120/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=118) | Arm B (N=121)
ALLERGIC REACTION (Immune system disorders) | 1 (2) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 2 (2)
AUTOIMMUNE DEFICIENCY SYNDROME (Immune system disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
FIBRILLATION ATRIAL (Cardiac disorders) | 2 (2) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
FAILURE HEART CONGESTIVE (Cardiac disorders) | 2 (2) | 2 (2)
HYPERTENSION (Cardiac disorders) | 0 (0) | 1 (2)
HYPOTENSION (Cardiac disorders) | 0 (0) | 2 (3)
MYOCARDIAL INFARCT (Cardiac disorders) | 0 (0) | 1 (1)
HEALING ABNORMAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HERNIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PYODERMA (SKIN INFECTION) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
KETOSIS (Endocrine disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (3)
BOWEL OBSTRUCTION (Gastrointestinal disorders) | 3 (3) | 1 (1)
BOWEL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLON OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLON ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 3 (3) | 7 (8)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FECAL IMPACTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL PERFORATION (NOS) (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (3) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (2) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 3 (3) | 0 (0)
INFECTION (Infections and infestations) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 4 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
FRACTURE BONE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DEPRESSION (Nervous system disorders) | 0 (0) | 1 (2)
HEADACHE (Nervous system disorders) | 1 (2) | 0 (0)
MENTAL DETERIORATION (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (2) | 0 (0)
PAIN (General disorders) | 1 (1) | 1 (2)
PERITONITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
PULMONARY EMBOLUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
ELECTROLYTE ABNORMALITY (Renal and urinary disorders) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
KIDNEY STONE (Renal and urinary disorders) | 0 (0) | 1 (2)
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 (0) | 1 (2)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 1 (2) | 1 (1)
THROMBOSIS (Vascular disorders) | 4 (4) | 7 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=118) | Arm B (N=121)
ALLERGIC REACTION (Immune system disorders) | 9 (13) | 4 (4)
HYPERSENSITIVITY (Immune system disorders) | 20 (42) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 45 (93) | 28 (57)
LEUKOPENIA (Blood and lymphatic system disorders) | 37 (142) | 26 (124)
NEUTROPENIA (Blood and lymphatic system disorders) | 49 (178) | 19 (87)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 42 (160) | 22 (66)
HYPERTENSION (Cardiac disorders) | 21 (32) | 15 (41)
HYPOTENSION (Cardiac disorders) | 1 (1) | 7 (8)
ASTHENIA (General disorders) | 13 (19) | 22 (31)
CHILLS (General disorders) | 9 (13) | 5 (5)
FATIGUE (General disorders) | 55 (115) | 40 (71)
FEVER (General disorders) | 15 (18) | 16 (20)
INSOMNIA (General disorders) | 16 (19) | 16 (17)
WEAKNESS GENERALIZED (General disorders) | 8 (9) | 9 (10)
WEIGHT LOSS (General disorders) | 19 (35) | 17 (22)
ACNE (Skin and subcutaneous tissue disorders) | 2 (3) | 34 (79)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (19) | 15 (16)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 21 (44)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 5 (10) | 9 (21)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (17)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (6) | 10 (19)
RASH (Skin and subcutaneous tissue disorders) | 17 (26) | 83 (168)
ABDOMINAL PAIN (Gastrointestinal disorders) | 26 (36) | 23 (25)
ANOREXIA (Gastrointestinal disorders) | 31 (51) | 29 (33)
CONSTIPATION (Gastrointestinal disorders) | 30 (42) | 36 (44)
DEHYDRATION (Gastrointestinal disorders) | 17 (22) | 8 (8)
DIARRHEA (Gastrointestinal disorders) | 53 (110) | 50 (105)
DYSGEUSIA (Gastrointestinal disorders) | 7 (10) | 5 (5)
DYSPHAGIA (Gastrointestinal disorders) | 7 (7) | 2 (2)
HEARTBURN (Gastrointestinal disorders) | 8 (9) | 2 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 8 (10)
MUCOSITIS NOS (Gastrointestinal disorders) | 14 (22) | 16 (26)
NAUSEA (Gastrointestinal disorders) | 59 (94) | 54 (103)
STOMATITIS (Gastrointestinal disorders) | 6 (7) | 19 (23)
VOMITING (Gastrointestinal disorders) | 32 (44) | 24 (31)
EPISTAXIS (General disorders) | 27 (30) | 18 (22)
INFECTION (Infections and infestations) | 8 (13) | 23 (27)
EDEMA (Blood and lymphatic system disorders) | 12 (17) | 9 (18)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 11 (20) | 7 (11)
HYPOCALCEMIA (Blood and lymphatic system disorders) | 6 (8) | 1 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 8 (13) | 13 (20)
HYPOMAGNESEMIA (Gastrointestinal disorders) | 10 (16) | 26 (27)
PROTEINURIA (Metabolism and nutrition disorders) | 10 (19) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (16) | 12 (16)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
ANXIETY (Psychiatric disorders) | 9 (9) | 6 (6)
DEPRESSION (Psychiatric disorders) | 7 (8) | 7 (7)
DIZZINESS (Nervous system disorders) | 14 (14) | 5 (7)
HEADACHE (Nervous system disorders) | 16 (20) | 16 (18)
NEUROPATHY (Nervous system disorders) | 68 (127) | 14 (25)
PARESTHESIA (Nervous system disorders) | 6 (13) | 0 (0)
TINGLING (Nervous system disorders) | 6 (7) | 1 (1)
PAIN (General disorders) | 20 (36) | 34 (51)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (14)
COUGHING (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 15 (18)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 18 (19)
INFECTION RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (7)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
URINARY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 10 (14)
THROMBOSIS (Vascular disorders) | 7 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes